CLINICAL TRIAL: NCT02221869
Title: A Multicenter Study of the Efficacy and Safety of Xyrem With an Open- Label Pharmacokinetic Evaluation and Safety Extension in Pediatric Subjects With Narcolepsy With Cataplexy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-005
Record Dates: First submitted 2014-07-28; First posted 2014-08-21 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Narcolepsy With Cataplexy
MeSH Terms: conditions — Narcolepsy | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xyrem (Experimental): Active Xyrem at a dose ≤9 g/night
  Interventions: Drug: Xyrem
- Xyrem Placebo (Placebo Comparator): Xyrem placebo at a volume and regimen equivalent to the stable dose of Xyrem.
  Interventions: Drug: Xyrem

INTERVENTIONS:
Drug: Xyrem

SUMMARY:
The purpose of this trial is to assess the efficacy and safety of Xyrem in pediatrics subjects with narcolepsy that includes cataplexy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 7-16 years at Visit 2 for subjects on Xyrem at study entry and at Visit 1.1 for Xyrem-naïve subjects (to ensure subjects are <18 years of age at the end of the study)
2. Have a primary diagnosis of narcolepsy with cataplexy that meets International Classification of Sleep Disorders (ICSD)-2 or ICSD-3 criteria, whichever was in effect at the time of the diagnosis or, with the permission of the Medical Monitor, completes a Multiple Sleep Latency Test (MSLT) during Screening to confirm the diagnosis of Type 1 narcolepsy by ICSD-3 criteria (i.e., the subject meets all other ICSD-3 criteria for Type 1 narcolepsy)
3. Have given documented assent indicating that he/she was aware of the investigational nature of the study and the required procedures and restrictions before participation in any protocol-related activities
4. Have parent(s)/guardian(s) who have given informed consent for his/her/their child's participation in the study
5. Be willing to spend the required number of nights (2 to 3) in a sleep laboratory for PSG evaluations
6. If currently treated with Xyrem, must have been taking unchanged doses (twice nightly dosing no higher than 9 g/night) of Xyrem, and stimulants, if applicable, for the treatment of narcolepsy symptoms for at least 2 months prior to screening

In addition to the above inclusion criteria, subjects participating in the PK evaluation must meet the following inclusion criteria:

7. Be willing to spend 2 additional nights in the clinic for PK evaluation

-

Exclusion Criteria:

1. Inability to understand assent or follow study instructions for any reason, in the opinion of the Investigator
2. Parent(s) or guardian(s) unable to comply with the requirements of the study for any reason, in the opinion of the Investigator
3. Other documented clinically significant condition (including an unstable medical condition, chronic disease other than narcolepsy with cataplexy, or history or presence of another neurological disorder) that might affect the subject's safety and/or interfere with the conduct of the study in the opinion of the Investigator
4. Treatment with benzodiazepines, non-benzodiazepine anxiolytics/ hypnotics/sedatives, neuroleptics, opioids, barbiturates, diclofenac, valproate, phenytoin, ethosuximide within 2 weeks prior to enrollment (discontinuation for the purpose of study enrollment is permitted only if considered safe by the Investigator and approved by the Medical Monitor)
5. Treatment with any other medications that have anticataplectic effect (e.g., serotonin-norepinephrine reuptake inhibitors [SNRIs], selective serotonin reuptake inhibitors [SSRIs], or tricyclic antidepressants [TCAs]) within 1 month before Screening
6. Unsafe for the subject to receive placebo treatment for 2 weeks, in the opinion of the Investigator

In addition to the above exclusion criteria, subjects participating in the PK evaluation must not demonstrate the following:

-

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (17):
  - Miller Children's Hospital - Long Beach, Long Beach, California
  - SDS Clinical Trials, Inc., Orange, California
  - Stanford Sleep Medicine Center, Redwood City, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The U-M Sleep Disorders Center, Ann Arbor, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Duke Children's Hospital, Durham, North Carolina
  - ARSM Research, LLC, Huntersville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - SleepMed of SC, Columbia, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - UT/LeBonheur Neuroscience Institute, Memphis, Tennessee
  - Todd Swick, MD, PA, Houston, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Hospital Robert Debre, Paris, France
- Dipartimento di Scienze Biomediche e Biomotorie, Bologna, Italy
- Sleep Wake Center SEIN Heemstede, Heemstede, North Holland, Netherlands

REFERENCES:
- [Derived] Dauvilliers Y, Lammers GJ, Lecendreux M, Maski K, Kansagra S, Black J, Parvataneni R, Chen A, Wang YG, Plazzi G. Effect of sodium oxybate on body mass index in pediatric patients with narcolepsy. J Clin Sleep Med. 2024 Mar 1;20(3):445-454. doi: 10.5664/jcsm.10912. PMID 37942930
- [Derived] Lecendreux M, Plazzi G, Dauvilliers Y, Rosen CL, Ruoff C, Black J, Parvataneni R, Guinta D, Wang YG, Mignot E. Long-term safety and maintenance of efficacy of sodium oxybate in the treatment of narcolepsy with cataplexy in pediatric patients. J Clin Sleep Med. 2022 Sep 1;18(9):2217-2227. doi: 10.5664/jcsm.10090. PMID 35689598
- [Derived] Wang YG, Menno D, Chen A, Steininger TL, Morris S, Black J, Profant J, Johns MW. Validation of the Epworth Sleepiness Scale for Children and Adolescents (ESS-CHAD) questionnaire in pediatric patients with narcolepsy with cataplexy aged 7-16 years. Sleep Med. 2022 Jan;89:78-84. doi: 10.1016/j.sleep.2021.11.003. Epub 2021 Nov 11. PMID 34920345
- [Derived] Plazzi G, Ruoff C, Lecendreux M, Dauvilliers Y, Rosen CL, Black J, Parvataneni R, Guinta D, Wang YG, Mignot E. Treatment of paediatric narcolepsy with sodium oxybate: a double-blind, placebo-controlled, randomised-withdrawal multicentre study and open-label investigation. Lancet Child Adolesc Health. 2018 Jul;2(7):483-494. doi: 10.1016/S2352-4642(18)30133-0. Epub 2018 May 21. PMID 30169321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 106 subjects were enrolled. Xyrem-naïve subjects (n=74) entered the Dose Titration Period (3 to 10 weeks). Xyrem-naïve and on Xyrem subjects (n= 99) entered the Stable Dose Period (2 to 3 weeks). 96 subjects then entered the Double-Blind Randomized Withdrawal Period (2 weeks). 95 subjects then entered the Open-label Safety Period (38 to 47 weeks).
Pre-assignment Details: Subjects aged 7-17 who were being treated with Xyrem or Xyrem naïve were eligible for the study. 63 subjects were randomized and 33 received open-label Xyrem during the Double-blind Treatment Period. 106 and 63 subjects comprised the Enrolled population and the Efficacy population respectively.
Groups:
- Randomized to Xyrem: Active Xyrem continued as a double-blind treatment at the stable dose taken and regimen taken in the prior 2 weeks.
- Randomized to Xyrem Placebo: Xyrem placebo was initiated as a double-blind treatment at a volume and regimen equivalent to the Xyrem dose taken in the prior 2 weeks.
- Open-label Xyrem: Subjects who were not randomized or continued to receive open-label Xyrem during the Double-blind Treatment Period.
Period: Overall Study
Arm/Group | Randomized to Xyrem | Randomized to Xyrem Placebo | Open-label Xyrem
Started | 31 | 32 | 43
Completed (Double-blind Period) | 30 | 32 | 33
Not Completed | 1 | 0 | 10

BASELINE CHARACTERISTICS:
Population: 106 subjects were enrolled. 63 subjects were randomized during the Double-blind Treatment Period. 106 subjects comprised the Enrolled population, and 63 subjects comprised the Efficacy population.
Groups:
- Enrolled Population: The Enrolled Population consists of all subjects who were dispensed study drug.
- Placebo (Efficacy Population): Xyrem placebo was initiated as a double-blind treatment at a volume and regimen equivalent to the Xyrem dose taken in the prior 2 weeks in the 2-week double-blind treatment period.
- Xyrem (Efficacy Population): Active Xyrem continued as a double-blind treatment at the stable dose taken and regimen taken in the prior 2 weeks in the 2-week double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Enrolled Population | Placebo (Efficacy Population) | Xyrem (Efficacy Population) | Total
Number analyzed (Participants) | 106 | 32 | 31 | 169
Age, Categorical [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Data analyzed separately for Enrolled and Efficacy populations
  Participants
    Enrolled Population: number analyzed (Participants) | 106 | 0 | 0 | 106
    Enrolled Population: <=18 years | 106 |  |  | 106
    Enrolled Population: Between 18 and 65 years | 0 |  |  | 0
    Enrolled Population: >=65 years | 0 |  |  | 0
    Efficacy Population: number analyzed (Participants) | 0 | 32 | 31 | 63
    Efficacy Population: <=18 years |  | 32 | 31 | 63
    Efficacy Population: Between 18 and 65 years |  | 0 | 0 | 0
    Efficacy Population: >=65 years |  | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Data analyzed separately for Enrolled and Efficacy populations
  Participants
    Enrolled Population: number analyzed (Participants) | 106 | 0 | 0 | 106
    Enrolled Population: Female | 43 | 0 |  | 43
    Enrolled Population: Male | 63 | 0 |  | 63
    Efficacy Population: number analyzed (Participants) | 0 | 32 | 31 | 63
    Efficacy Population: Female |  | 15 | 13 | 28
    Efficacy Population: Male |  | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Data analyzed separately for Enrolled and Efficacy populations
  Participants
    Enrolled Population: number analyzed (Participants) | 106 | 0 | 0 | 106
    Enrolled Population: Hispanic or Latino | 6 |  |  | 6
    Enrolled Population: Not Hispanic or Latino | 100 |  |  | 100
    Enrolled Population: Unknown or Not Reported | 0 |  |  | 0
    Efficacy Population: number analyzed (Participants) | 0 | 32 | 31 | 63
    Efficacy Population: Hispanic or Latino |  | 2 | 0 | 2
    Efficacy Population: Not Hispanic or Latino |  | 30 | 31 | 61
    Efficacy Population: Unknown or Not Reported |  | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Data reported for the Enrolled Population
  Participants
    Netherlands: number analyzed (Participants) | 106 | 0 | 0 | 106
    Netherlands | 8 | 0 | 0 | 8
    United States: number analyzed (Participants) | 106 | 0 | 0 | 106
    United States | 62 |  |  | 62
    Italy: number analyzed (Participants) | 106 | 0 | 0 | 106
    Italy | 25 |  |  | 25
    France: number analyzed (Participants) | 106 | 0 | 0 | 106
    France | 10 |  |  | 10
    Finland: number analyzed (Participants) | 106 | 0 | 0 | 106
    Finland | 1 |  |  | 1
Region of Enrollment [Number; unit: participants] — Population: Measure Analysis Population Description: Data reported for Efficacy Population
  participants
    Netherlands: number analyzed (Participants) | 0 | 32 | 31 | 63
    Netherlands |  | 3 | 2 | 5
    United States: number analyzed (Participants) | 0 | 32 | 31 | 63
    United States |  | 17 | 16 | 33
    Italy: number analyzed (Participants) | 0 | 32 | 31 | 63
    Italy |  | 9 | 9 | 18
    France: number analyzed (Participants) | 0 | 32 | 31 | 63
    France |  | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Number of Cataplexy Attacks
Description: Double-blind comparison of the change in weekly number of cataplexy attacks from the last 2 weeks of the Stable Dose Period to the 2 weeks of the Double-blind Treatment Period.
Time Frame: From the end of the Stable Dose Period to the end of the Double-blind Treatment Period (2 weeks)
Measure: Median (Inter-Quartile Range); unit: number of attacks
Groups:
- Xyrem: Active Xyrem continued as a double-blind treatment at the stable dose taken and regimen used in the prior 2 weeks.
- Xyrem Placebo: Xyrem placebo was initiated as a double-blind treatment at a volume and regimen equivalent to the Xyrem dose taken in the prior 2 weeks.
Arm/Group | Xyrem | Xyrem Placebo
Number analyzed (Participants) | 31 | 32
number of attacks | 0.27 [-1.00 to 2.50] | 12.71 [3.44 to 19.77]

2. Secondary Outcome: Clinical Global Impression of Change (CGIc) for Cataplexy Severity
Description: CGIc for cataplexy severity from the end of the Stable Dose Period to the end of the Double-blind Treatment Period.
  The CGIc is a 7-point scale ranging from "very much improved" to "very much worse." A score of 0 = no change, a score of 3 = very much improved, and a score of -3 = very much worse.
Time Frame: From the end of the Stable Dose Period to the end of the Double-blind Treatment Period (2 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xyrem | Xyrem Placebo
Number analyzed (Participants) | 29 | 32
score on a scale | -0.4 (1.12) | -1.5 (1.19)

3. Secondary Outcome: Change in the Epworth Sleepiness Scale (ESS) (CHAD) Score
Description: Change in the ESS (CHAD) score from the end of the Stable Dose Period to the end of the Double-blind Treatment Period.
  The ESS is a self-administered questionnaire with 8 questions. It provides a measure of a person's general level of daytime sleepiness, or their average sleep propensity in daily life. In the ESS for children and adolescents (CHAD), certain activities were modified. Each activity is scored on a scale ranging from 0-3, with 0 = would never fall asleep, and 3 = high chance of falling asleep. The total score ranges from 0-24, with a higher number representing an increased propensity for sleepiness.
Time Frame: From the end of the Stable Dose Period to the end of the Double-blind Treatment Period (2 weeks)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Xyrem | Xyrem Placebo
Number analyzed (Participants) | 30 | 31
score on a scale | 0.0 [-1.0 to 2.0] | 3.0 [1.0 to 5.0]

4. Secondary Outcome: CGIc for Narcolepsy Overall
Description: CGIc for narcolepsy overall from the end of the Stable Dose Period to the end of the Double-blind Treatment Period.
  The CGIc is a 7-point scale ranging from "very much improved" to "very much worse." A score of 0 = no change, a score of 3 = very much improved, and a score of -3 = very much worse.
Time Frame: From the end of the Stable Dose Period to the end of the Double-blind Treatment Period (2 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Xyrem | Xyrem Placebo
Number analyzed (Participants) | 29 | 32
score on a scale | -0.4 (0.95) | -1.4 (1.13)

5. Secondary Outcome: Change in Quality of Life (QoL; SF-10 Physical and Psychosocial Summary Score) From the End of the Stable Dose Period to the End of the Double-blind Treatment Period
Description: The SF-10 Health Survey for Children is a parent-completed survey that contains 10 questions adapted from the Child Health Questionnaire. The SF-10 is intended to produce physical and psychosocial health summary measures. Each of the 10 questions responses is scored with a point value from 1 to 6 (1 is the worst possible condition and 6 is the best possible condition). The SF-10 physical and psychosocial measures are scored such that higher scores indicate more favorable functioning.
  The questions and associated point values are separated into the Physical Health (PHS-10 domain) and Psychosocial Health (PSS-10 domain). The sums of the scores in each domain are standardized using the mean and standard deviation from a normal population (2006 sample). The standardized scores are transformed to norm based scoring (NBS) metric. Through NBS, scale scores are standardized to a mean of 50 and SD of 10 in the combined U.S. general population and clinical samples. NBS scores are reported
Time Frame: From the end of the Stable Dose Period to the end of the Double-blind Treatment Period (2 weeks)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Xyrem | Xyrem Placebo
Number analyzed (Participants) | 30 | 30
score on a scale
  SF-10 Physical Summary Score | 0 [-2.730 to 2.500] | 0 [-8.420 to 2.730]
  SF-10 Psychosocial Summary Score | 0 [-6.240 to 2.680] | -2.670 [-8.020 to 2.670]

ADVERSE EVENTS:
Time Frame: Safety data are provided through the 120 day update.
Description: The Safety Population included all subjects who took study drug, and consisted of 104 subjects. There are 2 subjects included in the Enrolled Population who were dispensed study drug, but did not take the medication and were subsequently discontinued. As a result, safety analyses focused on the 104 subjects in the Safety Population. Adverse events are reported by the Safety Population in order to capture adverse events occurring across all treatment periods.
Groups:
- Safety Population: Safety population who took study drug
- Randomized Placebo: Subjects assigned to the Randomized Placebo group during the Double-blind Treatment Period. Adverse events with onset on or after the first dose in the Double-blind Treatment Period and prior to the date of first dose in the Open-label Safety Period are presented.
Arm/Group | Safety Population | Randomized Placebo
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/32
Serious Adverse Events (participants affected / at risk) | 2/104 | 0/32
Other Adverse Events (participants affected / at risk) | 80/104 | 10/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=104) | Randomized Placebo (N=32)
Acute Psychosis (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=104) | Randomized Placebo (N=32)
Enuresis (Renal and urinary disorders) | 20 | 1
Nausea (Gastrointestinal disorders) | 20 | 0
Vomiting (Gastrointestinal disorders) | 19 | 0
Headache (Nervous system disorders) | 18 | 0
Weight decreased (Investigations) | 12 | 1
Decreased appetite (Metabolism and nutrition disorders) | 9 | 0
Nasopharyngitis (Infections and infestations) | 9 | 0
Upper respiratory tract infection (Infections and infestations) | 9 | 0
Dizziness (Nervous system disorders) | 8 | 0
Somnolence (Nervous system disorders) | 2 | 7
Cataplexy (Nervous system disorders) | 2 | 6
Sleep disorder (Psychiatric disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Study Protocol (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT02221869/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT02221869/SAP_001.pdf